CLINICAL TRIAL: NCT00913614
Title: Single Dose, Open Label Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Evaluation of Three Different Eplivanserin Doses in Children Aged 6-17 Years With Insomnia of Various Origins
Brief Title: Single Dose Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Evaluation of Eplivanserin in Children With Insomnia
Acronym: PKiDs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKD10491
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: insomnia pediatric safety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — SR 46349B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Age Group 6-11 year old - Dose level 1 (Experimental)
  Interventions: Drug: Eplivanserin (SR46349)
- Age Group 6-11 year old - Dose Level 2 (Experimental)
  Interventions: Drug: Eplivanserin (SR46349)
- Age Group 6-11 year old - Dose Level 3 (Experimental)
  Interventions: Drug: Eplivanserin (SR46349)
- Age Group 12-17 year old - Dose level 1 (Experimental)
  Interventions: Drug: Eplivanserin (SR46349)
- Age Group 12-17 year old - Dose level 2 (Experimental)
  Interventions: Drug: Eplivanserin (SR46349)
- Age Group 12-17 year old - Dose level 3 (Experimental)
  Interventions: Drug: Eplivanserin (SR46349)

INTERVENTIONS:
Drug: Eplivanserin (SR46349) — Oral administration

SUMMARY:
Given the potential age-related differences in safety, tolerability, pharmacokinetics, and differences in sleep architecture in young children versus adolescent versus adult, studies to identify the appropriate drug and dosage for children of all ages are essential in addressing this health problem that impacts the child and their family. The objective of this study is to evaluate the safety, pharmacokinetics and preliminary efficacy of eplivanserin.

Primary objective: to assess the safety and tolerability after administration of single ascending oral doses of eplivanserin to children aged 6-17 years with insomnia of various origins.

To assess the pharmacokinetics of eplivanserin (and active metabolite: SR141342) after administration of single ascending oral doses of eplivanserin to children aged 6-17 years with insomnia of various origins.

Secondary objective: to assess the effect of single ascending oral doses of eplivanserin on global sleep parameters and sleep architecture measured via polysomnography recordings in children aged 6-17 years old with insomnia of various origins.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of insomnia of various origins.
* Complaint of childhood insomnia as defined by repeated difficulty with sleep initiation or consolidation that occurs despite adequate age appropriate time and opportunity for sleep. The existence of sleep difficulty will be supported by statements from the child and/or the caregiver that sleep is not properly initiated or maintained.
* Written consent must be obtained from the parent/legal guardian.
* Written assent must be obtained from children of the appropriate age who are capable of giving assent as determined by parent/legal guardian.

Exclusion Criteria:

* The sleep disturbance must not be attributable to either the direct physiologic effect of a drug of abuse or misuse of a prescribed medication.
* Subject, if female of childbearing potential, which are unwilling to abstain from sexual intercourse or practice a double contraception method for the length of the study.
* Mental retardation.
* The presence of any untreated or uncompensated clinically significant renal, endocrine, hepatic, respiratory, cardiovascular, neurologic (excluding ADHD), hematologic, immunologic, cerebrovascular disease, or malignancy.
* Subjects with a history of any significant gastrointestinal disease.
* Presence of drug or alcohol abuse within one year before inclusion.
* Current history of substance abuse/dependence.
* Pregnant or breast-feeding.
* Use of any hypnotics/psychotropics, antihistamines, melatonin, herbal products, or other sleep aids including clonidine for initiation or maintenance of sleep within one week or five half lives (whichever is longer), prior to screening and unwillingness to discontinue them at the screening visit.
* Subject tested positive at screening or at baseline or at Day 1, on urine drug screen for drugs known to alter sleep (amphetamine/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates and alcohol).
* Inability to swallow a pill in similar size as the tablets to be administered for this study.
* Current or recent (<60 days) participation in another clinical trial receiving an investigational drug.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety in terms of adverse events, laboratory tests, vital signs, ECGs | Up to 12 days following single dose administration
Pharmacokinetics parameters | on Day 1, Day 2, Day 5, Day 7 and Day 10

SECONDARY OUTCOMES:
Global sleep parameters | Immediately following single dose administration
Sleep architecture | Immediately following single dose administration

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States